CLINICAL TRIAL: NCT06707389
Title: A Pilot Study of Autologous Blood Monocyte Vesicles for the Treatment of Sudden Deafness
Brief Title: Autologous Blood Monocyte Vesicles for the Treatment of Sudden Deafness
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2023-1250-02
Record Dates: First submitted 2024-07-11; First posted 2024-11-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Sudden Deafness; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden; Hearing Loss, Sensorineural | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control (Active Comparator): Intratympanic injection of methylprednisolone (methylprednisolone succinic acid for injection) at a dose of 40mg/mL, three times a week. 40mg of methylprednisolone was dissolved in 0.2 ml of lidocaine injection and 0.8 ml of sterilized injection water.
  Interventions: Drug: Methylprednisolone
- apoVs(lower dose) (Experimental): Intratympanic injection of autologous blood monocyte vesicles, three times a week. Autologous blood monocyte vesicles were extracted from 20 ml peripheral blood from patients and dissolved in 0.2 ml of lidocaine injection and 0.8 ml of sterilized injection water.
  Interventions: Biological: autologous blood monocyte vesicles (lower dose)
- apoVs(higher dose) (Experimental): Intratympanic injection of autologous blood monocyte vesicles, three times a week. Autologous blood monocyte vesicles were extracted from 50 ml peripheral blood from patients and dissolved in 0.2 ml of lidocaine injection and 0.8 ml of sterilized injection water.
  Interventions: Biological: autologous blood monocyte vesicles (higher dose)

INTERVENTIONS:
Biological: autologous blood monocyte vesicles (lower dose) — 20 ml peripheral venous blood was extracted from each patient, anticoagulated with heparin and diluted with PBS. Peripheral blood mononuclear cells were isolated by Ficoll stratified solution. Extracellular vesicles of mononuclear cells were extracted by gradient centrifugation (800g centrifugation at 4 ℃ for 10 minutes, then 2000g centrifugation at centrifuged at 4 ℃ for 10 minutes and then 16000g centrifugation at 4 ℃ for 30 minutes. The precipitate was taken as monocyte vesicle and stored in refrigerator at 4 ℃. For intratympanic injection, precipitate was dissolved in 0.2 ml of lidocaine and 0.8 ml of sterilized injection water. Intratympanic injection of apoVs was performed three times a week.
  Arms: apoVs(lower dose)
Drug: Methylprednisolone — 40mg of methylprednisolone was dissolved in 0.2 ml of lidocaine injection and 0.8 ml of sterilized injection water. Intratympanic injection of methylprednisolone was performed three times a week.
  Arms: control
Biological: autologous blood monocyte vesicles (higher dose) — 50 ml peripheral venous blood was extracted from each patient, anticoagulated with heparin and diluted with PBS. Peripheral blood mononuclear cells were isolated by Ficoll stratified solution. Extracellular vesicles of mononuclear cells were extracted by gradient centrifugation (800g centrifugation at 4 ℃ for 10 minutes, then 2000g centrifugation at centrifuged at 4 ℃ for 10 minutes and then 16000g centrifugation at 4 ℃ for 30 minutes. The precipitate was taken as monocyte vesicle and stored in refrigerator at 4 ℃. For intratympanic injection, precipitate was dissolved in 0.2 ml of lidocaine and 0.8 ml of sterilized injection water. Intratympanic injection of apoVs was performed three times a week.
  Arms: apoVs(higher dose)

SUMMARY:
Sudden deafness is a common emergency in otorhinolaryngology. As the etiology and mechanism of sudden deafness remains unknown, there is no specific treatment. Therefore, to explore new treatments for sudden deafness is a urgent and challenging problem. Extracellular vesicles therapy has been proved to be effective for several diseases. From our previous study, extracellular vesicles from mesenchymal stem cell can effectively improve noise-induced sensorineural deafness in mice. While mesenchymal stem cell therapy faces immune rejection in clinical use, the investigators use autologous blood monocyte vesicles to avoid immune rejection and guarantee patients' safety. In this interventional study, the investigators aimed to study the clinical effects and adverse reactions of autologous blood monocyte vesicle therapy in the treatment of sudden deafness. A total of 30 patients with severe or worse sudden deafness will enroll in this study and randomly assigned to 3 group, which are control group (Intratympanic glucocorticoid injection), lower-dose apoVs group (lower dose of Intratympanic monocyte vesicles injection) and higher-dose apoVs group (higher dose of Intratympanic monocyte vesicles injection). This study will further promote new treatment for sudden deafness and improve the quality of life and prognosis of patients with sudden deafness, especially those with severe or extremely severe deafness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65.
* Patients with severe and above unilateral hearing loss who meet the diagnostic criteria for sudden deafness.
* Patients who suffer sudden deafness within 3 weeks and do not receive intratympanic injection.
* Patients who fully understand the purpose and requirements of the trial, volunteer to participate in the clinical trial, sign a written informed consent, and is willing to complete the whole trial process according to the trial requirements.

Exclusion Criteria:

* Patients with conductive deafness and mixed deafness;
* Patients with other otologic diseases;
* Those who have doubts about the treatment plan or have obvious mental and psychological disorders;
* Patients with severe heart, lung, liver and kidney dysfunction;
* Patients with severe hematological diseases or tumors (especially those with acoustic neuromas);
* Those with positive HIV antibody, HBsAg, HCV antibody, or serological examination results for syphilis;
* Patients with a history of infection within 1 month prior to screening, requiring hospitalization and / or antibiotics, or currently using systemic hormones (corticosteroids), immunosuppressants or cytotoxicity;
* Patients with a history of immune system diseases or hematological system diseases;
* Patients with abnormal blood findings, such as abnormal number and morphology of red blood cells, white blood cells and platelets;
* Patients with severe or unstable cardiovascular, respiratory, liver, kidney, blood, endocrine, and central nervous system diseases;
* Women during lactation, pregnancy, or possibly pregnancy;
* Patients with contraindications or allergies to the treatment of this study;
* Those who have participated in any clinical drug trial in the past 3 months;
* Patients that the Investigator considers unsuitable to participate in the trial;
* Patients not suitable for tympanic injection therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Audiometry | 4 weeks after intervention.
  Pure tone audiometry.

SECONDARY OUTCOMES:
Audiometry | 1 week, 2 weeks after intervention
  Pure tone audiometry
THI scale | 1 week, 2 weeks, 4 weeks after intervention.
  THI (tinnitus handicap inventory) is one of the most widely used tinnitus self-rating scales in the world.It consists of three dimensions: functional, emotional and severity and effect of decreased tinnitus on patients' daily life. The THI score is totally 100 points. The more score participants get, the severer tinnitus symtoms they suffer from. According to the total score, paticipants were divided into five grades, Grade I (0-16, light) , Grade II (18-36, mild) , Grade III (38-56, moderate) , grade IV (58-76, severe) , grade V (78-100, catastrophic).
Tinnitus VAS | 1 week, 2 weeks, 4 weeks after intervention.
  The VAS(visual analogue scale) for subjective severity of tinnitus focuses on the subjective assessment of general sensation. The VAS has a scale score of 0 to 10, with 0 being completely unaffected and 10 being very severely affected.
SAS | 1 week, 2 weeks, 4 weeks after intervention.
  The SAS(Self-Rating Anxiety Scale) consists of 20 items which reflect the subjective and feeling of Anxiety. The more score paticipants get, the more anxiety they suffer. The SAS score can be divided into 4 levels: normal(less than 50 score), mild anxiety(50-59 score), moderate anxiety(60-69 score) and severe anxiety(more than 69 score).
Adverse Events | 1 week, 2 weeks, 4 weeks after intervention.
  Local adverse events include hearing loss, otitis media, and unperforation of tympanic membrane. Systemic adverse events include vital signs instability, new-onset anemia, liver and kidney dysfunction and so on. The severity of adverse events was graded according to the Common Adverse Event Evaluation Criteria (CTCAE) 5.0, Grade 1: mild; asymptomatic or mild; clinical or diagnostic only; treatment free. Grade 2: Moderate; requiring small, local, or non-invasive treatment; limited instrumental daily living activities comparable to age. Grade 3: serious or medically significant but not immediately life threatening; hospitalization or prolonged hospitalization; disability; limited activities of daily life. Grade 4: life-threatening; requiring urgent treatment. Grade 5: Death related to AEs.